CLINICAL TRIAL: NCT02214706
Title: Treatment of Port Wine Stains Using Pulsed Dye Laser, Erbium Yag Laser and Topical Sirolimus in an Open Label Pilot Study (POLAR).
Brief Title: Treatment of Port Wine Stains Using Pulsed Dye Laser, Erbium Yag Laser and Topical Sirolimus
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of efficacy / adverse events
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, M.B.A. van Doorn, MD, PhD, Erasmus Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EMC14022_POLAR
Record Dates: First submitted 2014-08-11; First posted 2014-08-12 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Port-Wine Stain
MeSH Terms: conditions — Port-Wine Stain | interventions — Sirolimus; Lasers, Solid-State; Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- sirolimus topical 40microgram/cm2 (Experimental): sirolimus topical 40microgram/cm2
  Interventions: Drug: Sirolimus
- Pulsed Dye Laser + Erbium yag + sirolimus (Experimental): Pulsed Dye Laser + Erbium yag laser + topical sirolimus
  Interventions: Drug: Sirolimus; Other: Erbium yag laser; Device: Pulsed Dye Laser
- Pulsed Dye Laser + topical sirolimus (Experimental): Pulsed Dye Laser + topical sirolimus
  Interventions: Drug: Sirolimus; Device: Pulsed Dye Laser
- Pulsed Dye Laser (Experimental): Pulsed Dye Laser
  Interventions: Device: Pulsed Dye Laser

INTERVENTIONS:
Drug: Sirolimus — sirolimus (40 µl) will be applied under occlusion, using van der Bend patch-test chambers (size: 1cm2), and left in situ for 7 days.
  Other Names: Rapamune
  Arms: Pulsed Dye Laser + Erbium yag + sirolimus; Pulsed Dye Laser + topical sirolimus; sirolimus topical 40microgram/cm2
Other: Erbium yag laser — Er:Yag laser ablation of the stratum corneum
  Arms: Pulsed Dye Laser + Erbium yag + sirolimus
Device: Pulsed Dye Laser
  Arms: Pulsed Dye Laser; Pulsed Dye Laser + Erbium yag + sirolimus; Pulsed Dye Laser + topical sirolimus

SUMMARY:
The purpose of this study is to improve the therapeutic outcome of laser therapy for port wine stains by using a combination treatment of the pulsed dye laser (PDL), erbium yag laser and topical sirolimus.

DETAILED DESCRIPTION:
In the first treatment period all patients will receive a total of five treatments with two week intervals. Every patient will receive the following four treatments (utilizing a template with separate squares of 1cm2): 1) PDL treatment followed by topical sirolimus application after Er:Yag laser ablation of the stratum corneum compared with 2) PDL treatment followed by topical sirolimus application without Er:Yag laser ablation of the stratum corneum, 3) PDL treatment only and 4) sirolimus application only. After the six months follow-up period, during the second treatment period, patients will receive an additional five treatments of the adjacent cosmetic unit of the treated part of the PWS, employing the most successful of the four treatment modalities as evaluated after the first treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided informed consent;
* Subject is ≥ 18 years of age at time of screening;
* Subject has an extra-facial homogenous Port Wine Stain (PWS);
* The PWS is large enough in size to fit one of the templates
* Subject has not received any laser treatment of the PWS in the last 3 months (in the treatment area);
* The PWS has a minimal erythema grading score of 3 (on a 4 point scale) in the opinion of the investigator;
* Screening blood safety values are within normal parameters or regarded as not clinically significant in the opinion of the investigator.

Exclusion Criteria:

* PWS with a nodular/hypertrophic component in the treatment area;
* PWS on cosmetically unacceptable locations in the opinion of the investigator;
* For women: pregnant or breast feeding during the treatment period;
* Women of child-bearing potential, unless they are using adequate contraceptive measures
* Subject is known to have immune deficiency, or is immune compromised
* Known allergy to sirolimus or other constituents of the study medication;
* Incapacitated subjects;
* Any medical or psychiatric condition which, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-07; Primary Completion 2016-01 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Percentage clearance assessed colorimetrically | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Martijn van Doorn, MD, Phd, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Greveling K, Prens EP, van Doorn MB. Treatment of port wine stains using Pulsed Dye Laser, Erbium YAG Laser, and topical rapamycin (sirolimus)-A randomized controlled trial. Lasers Surg Med. 2017 Jan;49(1):104-109. doi: 10.1002/lsm.22548. Epub 2016 Jun 20. PMID 27320685